CLINICAL TRIAL: NCT04910945
Title: Pilot Study for the Clinical Evaluation of Mechanical Coring to Achieve Directional Skin Tightening
Brief Title: Mechanical Coring to Achieve Directional Skin Tightening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI0620
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Skin Tightening; Healthy Volunteers
Keywords: Rhytides; Wrinkles; Loose Skin; Skin Laxity; Mechanical Coring; Robotic Coring; Skin Scarring; Scars; Stretch marks
MeSH Terms: conditions — Cutis Laxa; Cicatrix; Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Micro-coring treatment (Experimental)
  Interventions: Device: VENUS AIME (RoboCor)

INTERVENTIONS:
Device: VENUS AIME (RoboCor) — VENUS AIME is a micro-coring device of the skin that can potentially help to reduce visible skin scarring, improve skin laxity and reduce wrinkles.

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of mechanical coring for directional skin tightening. This study is a prospective, up to 3 center, multiple skin treatment area study of the safety and efficacy of mechanical coring with directional closure to achieve directional skin tightening.

DETAILED DESCRIPTION:
The study will evaluate the progress of up to 70 subjects after one treatment at up to 6 treatment areas on the body chosen from 2 on the neck (each treatment area approximately 1x3 cm), 2 on each underarm, 1 on each cheek, 2 on the abdomen, one on each thigh and 2 on the forehead area above the eyebrows (all approximately 6x4 cm). Subjects will be followed at 2, 5, 14, 28, 60, and 90 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects between 30 and 70 years of age.
2. Able to read, understand, and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of childbearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.
5. Subjects may have any Fitzpatrick skin type, however, no more than 35% of subjects may have Fitzpatrick skin type V or VI.

Exclusion Criteria:

1. Previous aesthetic (device and/or surgical) skin treatment in the treated areas (under arms and/or behind the ear) in the previous 6 months.
2. Fat, collagen, silicone, tattoos, body jewelry, that cannot be removed for the duration of treatment, and tegaderm/glue application or any other synthetic material in the treatment area.
3. History of keloid formation
4. Active smoker or having quit smoking in the last 3 months.
5. Active, chronic, or recurrent infection
6. Compromised immune and/or healing system (e.g. diabetes)
7. Hypersensitivity/allergy to analgesic agents, Betadine, tumescent, Benzoin Tincture, Tegaderm or tensioning tape that will be used in the study.
8. Co-morbid condition that could limit the ability to participate in the study or to comply with follow-up requirements.
9. Pregnant or breastfeeding
10. Any indication that may cause excessive bleeding, e.g., anticoagulants.
11. Carcinoma, melanoma, or any other cancerous condition in the last 6 months.
12. Allergy to adrenaline, epinephrine, or Tranexamic acid (TXA).
13. Currently or in the last 1-month part of another clinical study of an investigational drug and/or experimental medical device
14. Any issue that, at the discretion of the investigator would contra-indicate the subject's participation.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Cores Successfully Removed by Coring Device | 1 day
  Percentage of cores successfully removed by the coring device without manual removal.

SECONDARY OUTCOMES:
Downtime, as evaluated using the Subject Questionnaire | Up to Day 90 (end of study)
  Made of 8 questions asking if subject felt self-conscious, covered up the treatment area, avoided people, unable to perform normal activities, felt pain, discomfort or itchiness. For each, the subject may answer 1) Not at all, 2) Some of the time, or 3) Most of the time. A lower score indicates a better result.

OTHER OUTCOMES:
Treatment pain | Day 1
  Subject's assessment of discomfort and pain after treatments as measured by a VAS Pain Scale on 10 cm line. 0 cm being no pain/no discomfort and 10 cm being excruciating and unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, PhD, Study Director — Venus Concept
Locations (3):
- United States (3):
  - Berman Skin Institute, Los Altos, California
  - Le's Aesthetics, San Jose, California
  - DeNova Research, Chicago, Illinois